CLINICAL TRIAL: NCT02209233
Title: Effects of Massage on Post-operative Pain in Urologic Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 5140181
Record Dates: First submitted 2014-07-10; First posted 2014-08-05 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Postoperative Pain; Anxiety
MeSH Terms: conditions — Pain, Postoperative; Anxiety Disorders | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): If randomized to the control group, patients will not be receiving massage therapy.
- Massage Therapy (Experimental): If randomized to the intervention group, patients will receive massage therapy of the hand, arm, shoulder, and neck by the licensed massage therapist on duty. The massage will be given in a manner that is congruent with standard of care practices by the Heart and Surgical Hospital and the licensed massage therapist.
  Interventions: Other: Massage Therapy

INTERVENTIONS:
Other: Massage Therapy
  Arms: Massage Therapy

SUMMARY:
The purpose of this study is to determine the effect that receiving massage therapy post-operatively has on reducing perceived anxiety and pain in urology patients. Secondarily, the result of massage on patient satisfaction, length of hospital stay, and narcotic use will also be studied.

DETAILED DESCRIPTION:
Post-operative pain for Urology patients can be an anxiety-provoking and distressing recovery process. Massage therapy for post-operative pain has been shown to reduce pain and anxiety levels in various surgical patients however no study has assessed massage therapy effect on post-operative pain in patients who have gone through urological procedures.

This study will investigate the effects of hand massage interventions during the post-operative period of Urology patients. Perception of pain and anxiety levels will be assessed, as well as vital signs before and after massage therapy will be measured. These findings may lead to both subjective and objective improvements in patients undergoing urological surgeries and procedures.

ELIGIBILITY:
Inclusion Criteria:

* Urology patients over the age of 18 years old who are post-operative day 1 to post-operative day 4.

Exclusion Criteria:

* Given pain medication in the past hour

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain on the visual analogue scale score and survey | Baseline, 0-1 hour after intervention
Change from baseline in anxiety on the State Trait Anxiety Inventory (STAI) | Baseline, 0-1 hours after intervention

SECONDARY OUTCOMES:
Change from baseline in patient satisfaction on the Patient Satisfaction Questionnaire 18 (PSQ18) | Baseline, 0-1 hours after intervention
Length of hospital stay by chart review | From enrollment to time of discharge, an expected average of 7 days
Narcotic use (dosage, frequency, etc.) by chart review | Participants will be followed for the duration of hospital stay, an expected average of 1 week

CONTACTS AND LOCATIONS:
Overall Officials: D. Duane Baldwin, M.D., Principal Investigator — Loma Linda University Medical Center
Locations (1):
- Loma Linda University Heart and Surgical Hospital, Loma Linda, California, United States

REFERENCES:
- [Background] Julian LJ. Measures of anxiety: State-Trait Anxiety Inventory (STAI), Beck Anxiety Inventory (BAI), and Hospital Anxiety and Depression Scale-Anxiety (HADS-A). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S467-72. doi: 10.1002/acr.20561. No abstract available. PMID 22588767
- [Background] Stanley MA, Novy DM, Bourland SL, Beck JG, Averill PM. Assessing older adults with generalized anxiety: a replication and extension. Behav Res Ther. 2001 Feb;39(2):221-35. doi: 10.1016/s0005-7967(00)00030-9. PMID 11153975
- [Background] Collins SL, Moore RA, McQuay HJ. The visual analogue pain intensity scale: what is moderate pain in millimetres? Pain. 1997 Aug;72(1-2):95-7. doi: 10.1016/s0304-3959(97)00005-5. PMID 9272792
- [Background] Kelly AM. The minimum clinically significant difference in visual analogue scale pain score does not differ with severity of pain. Emerg Med J. 2001 May;18(3):205-7. doi: 10.1136/emj.18.3.205. PMID 11354213
- [Background] Reed MD, Van Nostran W. Assessing pain intensity with the visual analog scale: a plea for uniformity. J Clin Pharmacol. 2014 Mar;54(3):241-4. doi: 10.1002/jcph.250. Epub 2014 Jan 23. No abstract available. PMID 24374753
- [Background] Campeau MP, Gaboriault R, Drapeau M, Van Nguyen T, Roy I, Fortin B, Marois M, Nguyen-Tan PF. Impact of massage therapy on anxiety levels in patients undergoing radiation therapy: randomized controlled trial. J Soc Integr Oncol. 2007 Fall;5(4):133-8. doi: 10.2310/7200.2007.018. PMID 19087756
- [Background] Bagheri-Nesami M, Shorofi SA, Zargar N, Sohrabi M, Gholipour-Baradari A, Khalilian A. The effects of foot reflexology massage on anxiety in patients following coronary artery bypass graft surgery: a randomized controlled trial. Complement Ther Clin Pract. 2014 Feb;20(1):42-7. doi: 10.1016/j.ctcp.2013.10.006. Epub 2013 Oct 25. PMID 24439644
- [Background] Kim MS, Cho KS, Woo H, Kim JH. Effects of hand massage on anxiety in cataract surgery using local anesthesia. J Cataract Refract Surg. 2001 Jun;27(6):884-90. doi: 10.1016/s0886-3350(00)00730-6. PMID 11408136
- [Background] Braun LA, Stanguts C, Casanelia L, Spitzer O, Paul E, Vardaxis NJ, Rosenfeldt F. Massage therapy for cardiac surgery patients--a randomized trial. J Thorac Cardiovasc Surg. 2012 Dec;144(6):1453-9, 1459.e1. doi: 10.1016/j.jtcvs.2012.04.027. Epub 2012 Sep 7. PMID 22964355
- [Background] Babaee S, Shafiei Z, Sadeghi MM, Nik AY, Valiani M. Effectiveness of massage therapy on the mood of patients after open-heart surgery. Iran J Nurs Midwifery Res. 2012 Feb;17(2 Suppl 1):S120-4. PMID 23833593
- [Background] Cutshall SM, Wentworth LJ, Engen D, Sundt TM, Kelly RF, Bauer BA. Effect of massage therapy on pain, anxiety, and tension in cardiac surgical patients: a pilot study. Complement Ther Clin Pract. 2010 May;16(2):92-5. doi: 10.1016/j.ctcp.2009.10.006. Epub 2009 Nov 14. PMID 20347840
- [Background] Wang AT, Sundt TM 3rd, Cutshall SM, Bauer BA. Massage therapy after cardiac surgery. Semin Thorac Cardiovasc Surg. 2010 Autumn;22(3):225-9. doi: 10.1053/j.semtcvs.2010.10.005. PMID 21167456
- [Background] Buyukyilmaz F, Asti T. The effect of relaxation techniques and back massage on pain and anxiety in Turkish total hip or knee arthroplasty patients. Pain Manag Nurs. 2013 Sep;14(3):143-54. doi: 10.1016/j.pmn.2010.11.001. Epub 2011 Jan 28. PMID 23972865
- [Background] Ucuzal M, Kanan N. Foot massage: effectiveness on postoperative pain in breast surgery patients. Pain Manag Nurs. 2014 Jun;15(2):458-65. doi: 10.1016/j.pmn.2012.03.001. Epub 2012 Jun 20. PMID 24882025
- [Background] Wang HL, Keck JF. Foot and hand massage as an intervention for postoperative pain. Pain Manag Nurs. 2004 Jun;5(2):59-65. doi: 10.1016/j.pmn.2004.01.002. PMID 15297952
- [Background] Thayaparan AJ, Mahdi E. The Patient Satisfaction Questionnaire Short Form (PSQ-18) as an adaptable, reliable, and validated tool for use in various settings. Med Educ Online. 2013 Jul 23;18:21747. doi: 10.3402/meo.v18i0.21747. No abstract available. PMID 23883565